CLINICAL TRIAL: NCT05440929
Title: Evaluation of the Acceptability, Appropriateness, and Feasibility/Usability of a Metastatic Breast-cancer Specific Prognostic Calculator Among Clinicians
Status: Recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2207
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Breast Cancer; End of Life
Keywords: Metastatic Breast Cancer; Prognostic Tool; End of life; Clinicians; Prognosis; Qualitative Interview; Caregivers
MeSH Terms: conditions — Breast Neoplasms; Death

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinicans: Participants will include: physicians, nurse practitioners, physician assistants, and nurse navigators. Participants will be recruited from the UNC Medical Center breast oncology group as well as other practices identified by the Principal Investigator based on existing professional networks (referring physicians, other UNC oncology entities, collaborative groups).
  Interventions: Behavioral: Clinician Qualitative Interview

INTERVENTIONS:
Behavioral: Clinician Qualitative Interview — Interviews will be conducted by experienced qualitative researchers from the UNC Connected Health for Applications & Interventions (CHAI) Core. The interview will be conducted over the phone or secure videoconferencing. The interview will be conducted in a semi-structured fashion using an interview guide. However, because the purpose of this semi-structured qualitative interview study is to determine which themes participants identify as important, the exact content of each interview will differ, and the interview guide will be modified as additional interviews are conducted. Interviews will be audio recorded with concurrent notetaking by the interviewer.

SUMMARY:
I this qualitative study, Investigators will conduct semi-structured interviews with clinicians that are involved in the care of patients with breast cancer to evaluate the acceptability, appropriateness, and feasibility/usability of a metastatic breast cancer-specific prognostic tool. These interviews will be conducted by the UNC CHAI Core and will continue until thematic saturation (estimated 10 participants). The investigators will code the qualitative data using emerging themes, guided by a well-established implementation science theory, the Consolidated Framework for Implementation Research (CFIR). The information gained from these studies will inform an implementation approach to increase the usability and acceptability of a novel prognostic tool to assist oncologists in the prognosis of patients with metastatic breast cancer.

DETAILED DESCRIPTION:
If this study is successful, Investigators will implement an MBC-specific prognostic tool to help clinicians identify patients who are at high risk of death in the next 30 days. Based on the input from clinicians in this proposal, as well as additional qualitative studies with patients and families, Investigators will design an implementation protocol to inform how to use this tool in clinical practice. Rather than simply publishing a prognostic tool that may not be adopted into practice, this project aims to ensure successful implementation of an evidence-based tool into the routine care of patients with MBC. Doing so will serve as an important step towards identifying high-risk patients and connecting ort to ensure high-quality, patient-centered end-of-life care.

ELIGIBILITY:
Inclusion Criteria:

1. Verbal informed consent obtained to participate in the study.
2. Subject is willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.
3. Physician, nurse practitioner, physician assistant, or nurse navigator
4. At least 6 months of experience in the clinical care of patients with metastatic breast cancer in the United States.

Exclusion Criteria:

* Non-English Speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinician participants will include physicians, nurse practitioners, physician assistants, and nurse navigators. Participants will be recruited from the UNC Medical Center breast oncology group as well as other practices identified by the Principal Investigator based on existing professional networks (referring physicians, other UNC oncology entities, collaborative groups).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2027-08-10 (Estimated)

PRIMARY OUTCOMES:
Key barriers for use a metastatic breast cancer-specific prognostic tool | 12 months
  Study Investigators have developed a metastatic breast cancer (MBC)-specific prognostic calculator using the ASCO CancerLinQ Discovery database to help oncologists better estimate prognosis in MBC patients. Key barriers using this metastatic breast cancer-specific prognostic tool will be identified, through semi-structured qualitative interviews with oncology clinicians.
Key facilitators for use of a metastatic breast cancer-specific prognostic tool | 12 months
  Study Investigators have developed a metastatic breast cancer (MBC)-specific prognostic calculator using the ASCO CancerLinQ Discovery database to help oncologists better estimate prognosis in MBC patients. Key facilitators using this metastatic breast cancer-specific prognostic tool will be identified, through semi-structured qualitative interviews with oncology clinicians.

SECONDARY OUTCOMES:
Key barriers for discussion of prognosis between oncology clinicians and patients with metastatic breast cancer | 12 months
  Key barriers for discussion of prognosis between oncology clinicians and patients with metastatic breast cancer will be identified, through semi-structured qualitative interviews with oncology clinicians.
Key facilitators for discussion of prognosis between oncology clinicians and patients with metastatic breast cancer | 12 months
  Key facilitators for discussion of prognosis between oncology clinicians and patients with metastatic breast cancer will be identified, through semi-structured qualitative interviews with oncology clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Ray, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States